CLINICAL TRIAL: NCT01250769
Title: Evaluating the Effect of a Novel Interproximal Cleaning Device on Oral Health
Brief Title: Evaluating the Effect of Tooth Cleaning Devices on Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Oral Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRC-0703
Record Dates: First submitted 2010-05-05; First posted 2010-12-01 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-08

CONDITIONS: Dental Plaque
Keywords: dental; dentist; plaque; IP Cleaning
MeSH Terms: conditions — Dental Plaque; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Manual Toothbrush 1 (Active Comparator): Manual Toothbrush used for 1 minute twice a day
  Interventions: Device: Manual Toothbrush
- Manual Toothbrush 2 (Active Comparator): Manual Toothbrush used for 2 minutes twice a day
  Interventions: Device: Manual Toothbrush
- Manual Toothbrush + Interproximal Cleaning 1 (Experimental): Manual Toothbrush used twice a day for 2 minutes plus Interproximal Cleaning Device used once a day
  Interventions: Device: Manual Toothbrush; Device: Interproximal Cleaning Device
- Manual Toothbrush + Interproximal Cleaning 2 (Experimental): Manual Toothbrush used twice a day for 2 minutes plus Interproximal Cleaning Device used twice a day
  Interventions: Device: Manual Toothbrush; Device: Interproximal Cleaning Device

INTERVENTIONS:
Device: Manual Toothbrush — A standard size manual toothbrush to clean visible tooth surfaces
  Other Names: ADA Reference Toothbrush
Device: Interproximal Cleaning Device — An electronic device that combines water and air to clean between the teeth
  Other Names: Philips AirFloss
  Arms: Manual Toothbrush + Interproximal Cleaning 1; Manual Toothbrush + Interproximal Cleaning 2

SUMMARY:
This is a study to evaluate the safety and the efficacy of tooth and interproximal cleaning modalities on oral health.

ELIGIBILITY:
Inclusion Criteria:

* are in good/excellent health;
* are 18 - 70 years old;
* have a minimum of 20 natural teeth (excluding 3rd molars);
* have sufficient test sites;
* have ≥ 20 bleeding sites;
* are willing to participate and available for participation.

Exclusion Criteria:

* have systemic diseases such as Down's syndrome, or known AIDS/HIV;
* have insulin dependant Diabetes;
* are pregnant or nursing by subject report;
* have a cardiac pacemaker
* are undergoing or require extensive dental or orthodontic treatment;
* require antibiotic treatment for dental appointments;
* have heavy deposits of calculus;
* have severe gingivitis or periodontitis;
* have extensive crown or bridge work and/or rampant decay;
* currently use bleaching trays;
* have any oral or extraoral piercing on lips or in mouth;
* have a professional prophylaxis within 4 weeks of study;
* participation in a prior study ≤ 20 days;
* employed by a oral healthcare products company or research institution.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Jenkins, Study Director — POHC
Locations (1):
- University Park Research Center, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Started | 11 | 73 | 75 | 11
Day 14 | 11 | 72 | 74 | 11
Completed | 11 | 72 | 73 | 11
Not Completed | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2 | Total
Number analyzed (Participants) | 11 | 72 | 74 | 11 | 168
Age Continuous [Mean (Standard Deviation); unit: years] — 1 subject who discontinued prior to Day 14 is excluded from the Manual Toothbrush 2 group
  1 subject who discontinued prior to Day 14 is excluded from Manual Toothbrush + Interproximal Cleaning Device 1 group
  years | 38.5 (12.60) | 39.6 (11.60) | 39.6 (10.90) | 41.2 (12.80) | 39.6 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants] — 1 subject who discontinued prior to Day 14 is excluded from the Manual Toothbrush 2 group
  1 subject who discontinued prior to Day 14 is excluded from Manual Toothbrush + Interproximal Cleaning Device 1 group
  Participants
    Female | 8 | 48 | 48 | 8 | 112
    Male | 3 | 24 | 26 | 3 | 56

OUTCOME MEASURES:

1. Primary Outcome: Residual Protein Concentration
Description: Residual protein concentration of interproximal plaque samples
Time Frame: 14 days
Population: Analysis of efficacy data was performed using a modified intent-to-treat population (MITT). The MITT Population included all randomized subjects with both a baseline and endpoint evaluation. Missing data were not imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Number analyzed (Participants) | 11 | 72 | 73 | 11
ug/mL | 33.5 [28.9 to 38.2] | 28 [26.2 to 29.8] | 20.4 [18.6 to 22.2] | 20.2 [15.6 to 24.9]

2. Secondary Outcome: Residual Protein Concentration
Description: Residual protein concentration of interproximal plaque samples
Time Frame: 28 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Number analyzed (Participants) | 11 | 72 | 72 | 11
ug/mL | 39.7 [33.2 to 46.2] | 36.2 [33.7 to 38.7] | 33.6 [31.1 to 36.2] | 33.9 [27.4 to 40.3]

3. Secondary Outcome: Modified Gingival Index
Description: Gingival inflammation evaluation on an ordinal scale of 0 to 4 (0 is best ; 4 is worst)
Time Frame: 14 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Number analyzed (Participants) | 11 | 72 | 74 | 11
units on a scale | 1.45 [1.27 to 1.63] | 1.48 [1.41 to 1.55] | 1.26 [1.19 to 1.33] | 1.39 [1.21 to 1.57]

4. Secondary Outcome: Modified Gingival Index
Description: Gingival inflammation evaluation on an ordinal scale of 0 to 4 (0 is best ; 4 is worst)
Time Frame: 28 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Number analyzed (Participants) | 11 | 72 | 73 | 11
units on a scale | 1.35 [1.18 to 1.52] | 1.44 [1.38 to 1.51] | 1.23 [1.17 to 1.3] | 1.41 [1.24 to 1.58]

5. Secondary Outcome: Gingival Bleeding Index
Description: Gingival bleeding evaluation using an ordinal scale of 0 to 3; (0 is best; 3 is worst)
Time Frame: 14 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Number analyzed (Participants) | 11 | 72 | 74 | 11
units on a scale | 0.36 [0.28 to 0.43] | 0.26 [0.23 to 0.29] | 0.18 [0.15 to 0.21] | 0.19 [0.12 to 0.27]

6. Secondary Outcome: Gingival Bleeding Index
Description: Gingival bleeding evaluation using a ordinal scale of 0 to 3; (0 is best; 3 is worst)
Time Frame: 28 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Number analyzed (Participants) | 11 | 72 | 73 | 11
units on a scale | 0.3 [0.23 to 0.38] | 0.26 [0.23 to 0.29] | 0.16 [0.13 to 0.19] | 0.2 [0.12 to 0.27]

ADVERSE EVENTS:
Arm/Group | Manual Toothbrush 1 | Manual Toothbrush 2 | Manual Toothbrush + Interproximal Cleaning 1 | Manual Toothbrush + Interproximal Cleaning 2
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/73 | 1/75 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/73 | 0/75 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Toothbrush 1 (N=11) | Manual Toothbrush 2 (N=73) | Manual Toothbrush + Interproximal Cleaning 1 (N=75) | Manual Toothbrush + Interproximal Cleaning 2 (N=11)
Left forearm deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Assessed by the PI as definitely not related to the investigational product. SAE outcome was recovered/resolved.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Toothbrush 1 (N=11) | Manual Toothbrush 2 (N=73) | Manual Toothbrush + Interproximal Cleaning 1 (N=75) | Manual Toothbrush + Interproximal Cleaning 2 (N=11)
Apthous ulcer above tooth #7 on attached gingiva (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Philips shall have the final authority to determine whether or not to publish study results.